CLINICAL TRIAL: NCT03192982
Title: Impact on Expected Post-operative Complications With Impulsive Compression of Vein Complexes in Foot of Patients Operated on With In-situ Bypass for Acute/Chronic Leg Ischemia
Brief Title: Post-operative Complication, Impulsive Compression, in Situ Bypass
Acronym: 50506
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kolding Sygehus (Other)
Responsible Party: Principal Investigator, Hans Ravn, Principal Investigator, Vejle Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Impulsive compression i insitu
Record Dates: First submitted 2017-05-29; First posted 2017-06-20 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Compresion Therapy; Post-operative Edema; Wound Complication; Ischemia Limb; Quality of Life

STUDY DESIGN:
Intervention Model Description: Randomized prospective study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Foot pump (A-V Impulse, 6000 Series) (Experimental): In OR before operation starts randomized to foot pump treatment post operative. Pump placed on foot immediately after operation is finished. Foot pump will be left on foot until full mobilization is reached
  Interventions: Device: A-V impulse 6000 Series
- Standard treatment (compression) (Active Comparator): In OR before operation starts randomized to standart treatment for edema after in situ bypass.
  Short-stretch bandage from toes and up yo the upper thigh 40 mm Hg
  Interventions: Device: Standard treatment (compression)

INTERVENTIONS:
Device: A-V impulse 6000 Series — foot pad and pump
  Arms: Foot pump (A-V Impulse, 6000 Series)
Device: Standard treatment (compression) — Short-stretch bandage from toes and up yo the upper thigh 40 mm Hg
  Arms: Standard treatment (compression)

SUMMARY:
To investigate whether compression therapy with foot pump reduce post-operative edema, facilitate wound healing of operation wounds, promote healing of ischemic ulcers and shorten hospitalization, increase and improve the patient's subjective quality of life faster

DETAILED DESCRIPTION:
Impact on expected post-operative complications with impulsive compression of vein complexes in foot of patient operated on with insitu bypass for acute/chronic leg ischemia.

Purpose/aim:

To investigate whether compression therapy with foot pump reduce post-operative edema, facilitate wound healing of the operation wounds, promote healing of ischemic ulcers and shorten hospitalization, increase and improve the patient's subjective quality of life faster.

Background:

Insitu bypass to the lower extremity are the standard operation choice on patients with critical leg ischemia. Approximately 18% of patients wound problems, which prolong their hospitalization time and convalescence. One of the reasons for wound problems is swelling, which occurs in connection with the legs process of revascularization (angiogenesis). One can expect that the leg, 10 cm below the patella will undergo swelling with approximately 6-8% during the first day, and up to 8-10% after four days in connection with the inset bypass surgery. Early mobilization can prevent the swelling to become too pronounced. By mobilizing you stimulate the natural venous pump in the leg. Patients are often hard to mobilize in an early stage due to the wound and age. Stimulation of the venous plexus in the arch of the foot has in other categories of patients shown to reduce swellings of leg and thrombosis risk in patients undergoing orthopedic surgery on the lower extremities .

There is no description of treatment of Vascular surgical patients with foot pump to be found in literature.

The patient's subjective quality of life is often impaired in relation to the above mentioned surgical treatment. A quicker recovery can be compatible with rapidly regained quality of life.

There is no analysis or meta Cochrane reviews in this field.

Plan and material:

- Procedure: Patients follow the normal procedure in the department in terms of insitu bypass.

Asked in the outpatient's clinic at visit for preparation for the operation.

- Method:

Time schedule for measuring assessing symptoms as pain, edema and swelling:

Measuring the leg swelling

1. The night before the operation.
2. The day after the operation.
3. Day 4 and the day of patient discharge.
4. Day 30 (control in our open clinic for control of the operation results).

   The measure procedure will be as follows:

   The circumference of the leg will be measured at 10 cm below the distal part of the patellae. In the same procedure pain by the Visual analogue scale (VAS) will evaluated and edema at the ankle in the same leg by digital pulpal pressure on the skin. The r reaction will be noted (fast recovery or slow) the depth of the dimple will be noted.

   Operation is planned.

   Post operation, foot pump is placed on foot, according to randomization. Pump must be placed on foot immediately after arrival to ICU. Foot pump will be left on foot until full mobilization is reached. The control group follows the department's ordinary post-operative routines for inset bypass, i.e. compression stockings or short-stretch bandage.

   The compression stocking is a TED stocking with 18 mmHg pressure at the ankle and short-stretch bandage is a padded bandage that stretch from the toes and up to the upper thigh with a 40 mmHg pressure.

   Time for full mobilization is recorded in all patients.

   Reoperations is noted.

   Toe pressure is measured at inclusion, immediately post-op and at discharge.

   Time for discharge is noted.

   Para clinical factors to be examined.

   Duplex study of reverse flow in the deep veins associated with standard duplex study of AV fistulas post-operatively.

   Quality of life questionnaire (vascu Qol)

   EQ-5D baseline + 6-month
   * Risks, side effects and disadvantages:

   The foot pump treatment is non-invasive. Patients bear no ache nor pain in connection with the treatment method. The pump is used in other European countries on an empirical basis and CE mark.

   Duplex study is done as routine examinations in the department and is non-invasive.

   The side effects and risks of pump therapy can be considered as insignificant.
   * Patient integrity:

   The project reported to the data monitoring via the regions" paraplyanmelselse" to the data inspectorate.

   The law on treatment of personal data will be respected.
   * Data application sheet:

   A data application sheet will be created for all the included patients. The information will be fed into the database for analysis. Usernames and passwords will be created for login for all trial related personnel.

   - Publication: The results of the study will be presented at national and international meetings and conventions. The end result will be published in an international magazine.

   - Ethical considerations: Wound complications associated with vascular surgery is a major problem for both patients and vascular surgeons. All that is possible to bring the infection rate down is good for patients and hospital systems. If we simultaneously can shorten the hospitalization time and improve the quality of life for patients, it will mean that we have accomplishment. This study is a win-win project without inflicting the trial subjects no significant risks or side effects. For research and surgical discipline, it can be of great importance to show the advantage with the foot pump treatment in a study. And thereby awaken the interest in foot pumps among other medical specialities.

   - Informed consent: Patients with critical leg ischemia, where there are taken a decision on inset bypass, is offered to participate in the trial by ambulatory visit. There will be a sheet with written information handed out and the patients will also receive information orally about the trial. The patient now has the option for consideration until the randomization will happen at admission to operation. The oral information will be given by the research nurse and study physician. The patient and Doctor/nurse call on a study room in the outpatient clinic at Department of Vascular surgery, Hospital Lillebaelt, Denmark.. The patient is given the written information to take home for reading and have the opportunity to have an observer present at the hospital where the patient must submit a statement of participation in the study. The tome between ambulatory visit and hospitalization in usually seven to 14 days depending on the severity of the patient's ischemia.

   - Patient Insurance: The subject is covered by the patient compensation scheme in the region of southern Denmark.

ELIGIBILITY:
Inclusion Criteria:

Patients who need an insitu bypass from Common Femoral Artery to Popliteal AK/BK or crural Artery

Exclusion Criteria:

Ischemic wound that are located in such manner that compression of the foot is not possible. Former deep vein trombosis (DVT) or symptomatic post thrombotic syndrome (PTS) We only include patients without any connections to other studies-

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-02-08 (Actual); Primary Completion 2022-11-28 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Reduction of wound complications in the foot pump group | From randomization until 12 month examination (individual finish examination)
  reduction from 18% to 14 %.Inspection of the operated leg at day 2 and 4 and at discharging. After discharging at 30 days, 6 month and one year.More frequent inspections can be necessary depending on the situation and the condition of the patient.
  Inspection of secretion from the operations cicatrices, necrosis and diastasis of the wounds, signs of infections, hematoma subcutaneously in the operation area, edema, temperature and color of the skin

SECONDARY OUTCOMES:
Reduction of leg edema 50%, | 5 to 30 days
  10 cm below the patella on the operated leg three days post-operation in patients treated with impulsive compression in comparison to non-treated.
Time to mobilization in pump treated patients | 1 to 7 days
  Patient can get out of bed and go to the toilet.
Length of stay in hospital | 10 to 14 Days

CONTACTS AND LOCATIONS:
Overall Officials: Hans Ravn, MD PhD, Study Chair — Vejle Hospital
Locations (1):
- Hans Ravn, Kolding, Denmark

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Klit T, Dahl M, Houlind KC, Ravn H. Effect of Impulsive Compression Treatment on Postoperative Complications After Open Peripheral Vascular Revascularization (In Situ): Protocol for a Randomized Control Trial. JMIR Res Protoc. 2018 Feb 20;7(2):e58. doi: 10.2196/resprot.8799. PMID 29463493